CLINICAL TRIAL: NCT04424511
Title: LAKANA , a Cluster-randomized, Double-blinded, Parallel Group, Controlled Trial, Testing the Effects of Mass Drug Administration of Azithromycin on Mortality and Other Outcomes Among 1-11 Month Old Infants in Rural Mali.
Brief Title: Effects of Mass Drug Administration of Azithromycin on Mortality and Other Outcomes Among 1-11 Month Old Infants in Mali
Acronym: LAKANA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tampere University (Other)
Collaborators: Center for Vaccine Development CVD-Mali, Bamako, Mali (Unknown); University College London Hospitals (Other); Tro Da Ltd, UK (Unknown); Duke-NUS Graduate Medical School (Other); Bill and Melinda Gates Foundation (Other); Pfizer Inc. (Provider of study drugs) (Unknown)
Responsible Party: Principal Investigator, Per Ashorn, MD, PhD, Professor of Pediatrics, Tampere University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAKANA trial; INV-003354 (Other Grant/Funding Number: Bill and Melinda Gates Foundation)
Record Dates: First submitted 2020-05-22; First posted 2020-06-11 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Mortality
Keywords: Mass Drug Administration; Azithromycin; Infant and Child Mortality; Infant and Child health; Infant and Child growth; Infant and Child morbidity; Antimicrobial Resistance; Feasibility; Acceptability; Safety; Cost; Inflammation; Infection
MeSH Terms: conditions — Inflammation; Infections | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: LAKANA is a cluster-randomized, placebo-controlled, double-blinded, parallel-group, three-arm clinical trial, with adaptive design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigators will utilize a matching placebo to mask study arm allocation. All children aged 1-11 months in all study communities will be offered biannual or quarterly azithromycin or placebo distribution in an identical fashion. Placebo will be identical to azithromycin in appearance, taste, odor, and packaging. The interventions will be coded only with a letter code.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Placebo Comparator): Placebo mixture will be administered as a single dose in oral suspension form for children 1-11 months of age:
  1. Single-dose of 0.5 ml / kg child weight
  2. Participating households within villages allocated to this group will be visited quarterly (at 3-month intervals), for nine times. At the first eight of these visits, 1-11 month old eligible infants, for whom there is a consent for study drug provision, will be weighed and given a single dose of placebo mixture.
  Interventions: Drug: Placebo
- Azithromycin-biannually (Azi-biannual) (Active Comparator): Azithromycin or placebo will be administered as a single dose in oral suspension form for children 1-11 months of age:
  1. Single-dose of 0.5 ml / kg child weight
  2. Participating households within villages allocated to this group will be visited quarterly (at 3-month intervals), for nine times. At the first eight of these visits, 1-11 month old eligible infants, for whom there is a consent for study drug provision, will be weighed and given a single dose of study drug.
  3. Azithromycin will be given at quarterly visits between January and June, and Placebo mixture will be given at quarterly visits between July and December. Azithromycin dose will be 20 mg / kg.
  Interventions: Drug: Placebo; Drug: Azithromycin
- Azithromycin-quarterly (Active Comparator): Azithromycin will be administered as a single dose in oral suspension form for children 1-11 months of age:
  1. Single-dose of 0.5 ml (20 mg) / kg child weight.
  2. Participating households within villages allocated to this group will be visited quarterly (at 3-month intervals), for nine times. At the first eight of these visits, 1-11 month old eligible infants, for whom there is a consent for study drug provision, will be weighed and given a single dose of azithromycin.
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Placebo — Placebo mixture will be administered as a single dose in oral suspension form for children 1-11 months of age. Weight-based dosing will be used: single-dose of 0.5 ml / kg child weight.
  Arms: Azithromycin-biannually (Azi-biannual); Control
Drug: Azithromycin — Azithromycin will be administered as a single dose in oral suspension form for children 1-11 months of age. Weight-based dosing will be used: single-dose of 0.5 ml (20 mg) / kg child weight.
  Arms: Azithromycin-biannually (Azi-biannual); Azithromycin-quarterly

SUMMARY:
The LAKANA trial will assess the impact on mortality and other health outcomes of quarterly and biannual azithromycin mass drug administration (MDA) when delivered to 1-11-month (29-364 days) old infants in a high-mortality setting where malaria is holoendemic but there is also a functioning seasonal malaria chemoprevention (SMC) program in place. The long-term goal is to more precisely define the role of mass azithromycin treatments as an intervention for reducing childhood mortality, and to determine the most effective treatment regimen. The main study hypotheses in terms of mortality effect are: i) Biannual azithromycin MDA to 1-11 month old infants reduces their mortality, ii) Quarterly azithromycin MDA to 1-11 month old infants reduces their mortality, iii) Quarterly azithromycin MDA has a bigger mortality effect than biannual MDA.

DETAILED DESCRIPTION:
Mass drug administration (MDA) of azithromycin has been shown to reduce under-5 mortality in some but not all sub-Saharan African settings. Because of the observed heterogeneity and possible effect modification by SMC or other co-interventions, further trials in new settings are needed in order to make evidence-based public health recommendations about the use of this treatment. The objectives of the LAKANA trial are:

* To evaluate the impact of two azithromycin MDA regimens on infant mortality and other health outcomes, when provided in a rural West-African high-mortality context with an ongoing seasonal malaria chemoprevention program.
* To evaluate the effect of alternative MDA frequencies on antimicrobial resistance (AMR) and host microbiota composition.
* To test hypotheses that azithromycin MDA eliminates malaria parasitaemia and reduces systemic and intestinal inflammation in asymptomatic children and to collect and store biological samples for assessing other possible mechanisms of azithromycin effect.
* To investigate the feasibility of alternative azithromycin MDA strategies, including economic analysis.

The LAKANA trial will be conducted in 1151 villages from 7-10 health districts in the Kayes, Kita and Koulikoro regions of Mali. LAKANA is a cluster-randomized, placebo-controlled, double-blinded, parallel-group, three-arm clinical trial, with adaptive design. Participating villages will be randomly allocated to three different intervention groups in a ratio of 3 : 2 : 4 (control : azithromycin quarterly : azithromycin biannually). Within each participating village, consenting households will be visited quarterly (at 3-month intervals), nine times. At the first eight of these visits, 1-11-month-old eligible infants (age 29-364 days), for whom there is a consent for study drug provision, will be given a single dose of study drug (azithromycin mixture or respective placebo mixture).

Mortality and serious adverse events (SAEs) data will be collected, and mortality-related questions answered using data from all the included 1151 villages. Mixed-effect Poisson regression model will be used to estimate the intervention effects on mortality, with random intercepts for the clusters. The investigators will explore effect modification by testing for interaction between the MDA intervention and the following variables:

* Age at the time of the MDA
* Sex of the child
* Weight-for-age
* Seasonality: rainy season vs non-rainy season at the time of the MDA
* SMC given to the child within 3 months before an MDA
* Order of MDA in the village
* District of residence
* Distance from the nearest health facility (in km)
* Household asset index
* Water, Sanitation, and Hygiene (WASH) index
* National outreach strategy category (standard/advanced)

The investigators will address the other study questions using a smaller separate secondary sample of 59 villages located around four selected health centers close to the city of Kita and a similar number of villages closer to Bamako, i.e. in Koulikoro or Kati (tertiary sample).

ELIGIBILITY:
Inclusion Criteria:

On a cluster (village) level:

1. Location within Kayes, Kita, or Koulikoro region of Mali
2. Considered accessible and safe by the local health authorities and research team
3. Considered non-urban by the local health authorities and research team
4. Permission from community leadership

On a household level (for trial enrollment):

1. Location within a cluster that is included in the study
2. Verbal consent from a head of household or an adult authorized by her / him

On a child level (for receiving study medication):

1. Residence in a household enrolled in the trial
2. Age between 29 and 364 days
3. Verbal consent from at least one caregiver

Exclusion Criteria:

On child level (for not receiving study medication):

1. Weight below 3.0 kg
2. Known allergy to macrolides, as judged by a caregiver report of the infant experiencing an adverse reaction after oral ingestion of medication, which was deemed likely to be a macrolide by the interviewing data collector.

Ages: 29 Days to 364 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 149201 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | 3-month time interval (total of 8 intervals per cluster)
  Mortality rate (deaths per 1,000 years at risk) among children 1-11 months of age.

SECONDARY OUTCOMES:
Morbidity | 3-month time interval (total of 8 intervals per cluster)
  Morbidity (14-day period prevalence of fever with respiratory symptoms (ARI), fever without respiratory symptoms (malaria), and diarrhea) in children aged 4-14 months assessed in each participating cluster (village) from the secondary outcome sample.
Length-for-age Z-score | 3-month time interval (total of 3 intervals per cluster)
  Length-for-age Z-score in 6-8 and 12-14 months old children from the secondary outcome sample. Length measures will be taken at 15, 18, 21, and 24 months after the enrollment of the village into the trial. Length-for-age Z-score will be calculated using the WHO Child Growth Standards.
Length | 3-month time interval (total of 3 intervals per cluster)
  Attained length in cm in 6-8 and 12-14 months old children from the secondary outcome sample. Length measures will be taken at 15, 18, 21, and 24 months after the enrollment of the village into the trial.
Weight | 3-month time interval (total of 3 intervals per cluster)
  Attained weight in grams in 6-8 and 12-14 months old children from the secondary outcome sample. Weight measures will be taken at 15, 18, 21, and 24 months after the enrollment of the village into the trial.
Weight-for age Z-score | 3-month time interval (total of 3 intervals per cluster)
  Weight-for age Z-score in 6-8 and 12-14 months old children from the secondary outcome sample. Weight measures will be taken at 15, 18, 21, and 24 months after the enrollment of the village into the trial. Weight-for-age Z-score will be calculated using the WHO Child Growth Standards.
Weight-for-length Z-score | 3-month time interval (total of 3 intervals per cluster)
  Weight-for-length Z-score in 6-8 and 12-14 months old children from the secondary outcome sample. Length and weight measures will be taken at 15, 18, 21, and 24 months after the enrollment of the village into the trial. Weight-for-length Z score will be calculated using the WHO Child Growth Standards.
Mid-upper arm circumference | 3-month time interval (total of 3 intervals per cluster)
  Mid-upper arm circumference in 6-8 and 12-14 months old children from the secondary outcome sample. Measures will be taken at 15, 18, 21, and 24 months after the enrollment of the village into the trial.
Percentage of moderate or severe stunting | 3-month time interval (total of 3 intervals per cluster)
  Percentage of moderate or severe stunting (length-for-age Z-score < -2 / -3) in 6-8 and 12-14 months old children from the secondary outcome sample.
Percentage of moderate or severe wasting | 3-month time interval (total of 3 intervals per cluster)
  Percentage of moderate or severe wasting (Weight-for-length Z-score < -2 / -3) in 6-8 and 12-14 months old children from the secondary outcome sample.
Percentage of moderate or severe Underweight | 3-month time interval (total of 3 intervals per cluster)
  Percentage of moderate or severe Underweight (Weight-for-age Z-score < -2 / -3) in 6-8 and 12-14 months old children from the secondary outcome sample.
Prevalence of phenotypic and genotypic macrolide resistance | 12-month time interval (total of 3 intervals per cluster)
  prevalence of phenotypic azithromycin resistance among S. pneumoniae or E. coli strains isolated from 4-14-month-old children, who have received 1-4 rounds of azithromycin MDA
Prevalence of phenotypic and genotypic macrolide resistance | 12-month time interval (total of 3 intervals per cluster)
  prevalence of phenotypic azithromycin resistance among S. pneumoniae or E. coli strains isolated from 49-59-month-old children, who live in the same Malian communities but have not received azithromycin MDA
Prevalence of phenotypic and genotypic macrolide resistance | 12-month time interval (total of 3 intervals per cluster)
  prevalence of phenotypic azithromycin resistance among S. pneumoniae or E. coli strains isolated from 15-26-month-old children, who have received 1-4 rounds of azithromycin MDA and live in a village that stopped azithromycin MDA 1 year before
Prevalence of phenotypic and genotypic macrolide resistance | 12-month time interval (total of 3 intervals per cluster)
  prevalence of phenotypic azithromycin resistance among S. pneumoniae or E. coli strains isolated from 24-35-month-old children, who have received 1-4 rounds of azithromycin MDA 1 year before and who live in a village that continued azithromycin MDA
Prevalence of phenotypic and genotypic AMR resistance to other "ACCESS" group antibiotics | 12-month time interval (total of 3 intervals per cluster)
  Prevalence of phenotypic and genotypic AMR against other antibiotics categorised by the World Health Organization (WHO) into "ACCESS" group, among azithromycin-resistant E. coli strains isolated from stool samples or azithromycin-resistant S. pneumoniae strains isolated from nasopharyngeal swabs (secondary outcome sample).
Blood C-reactive protein concentration | Biological samples taken before and 14 days after the fourth MDA round, 9 months after village enrollment.
  Biological samples taken from 4-11 months old infants to assess effect of azithromycin MDA on systemic inflammation (blood C-reactive protein concentration) (secondary outcome sample).
Blood malaria parasitemia and hemoglobin concentration | Biological samples taken before and 14 days after the fourth MDA round, 9 months after village enrollment.
  Biological samples taken from 4-11 months old infants to assess effect of azithromycin MDA on malaria prevalence and blood hemoglobin concentration (secondary outcome sample).
Fecal neopterin, myeloperoxidase, and alpha-1-antitrypsin concentrations | Biological samples taken before and 14 days after the fourth MDA round, 9 months after village enrollment.
  Biological samples taken from 4-11 months old infants to assess effect of azithromycin MDA on intestinal inflammation and function (secondary outcome sample).
Incidence of Adverse events | 3-month time interval
  Incidence of adverse events within 14 days of study drug administration. Data collected from 4-11 months old infants at 9 months after enrollment (secondary outcome sample).
Incidence of Serious Adverse events | within 14 days after MDA round.
  Incidence of serious adverse events (Death, life-threatening event, hospitalization, and other serious events as judged by a study physician) within 14 days of study drug administration, among 1-11 months old infants.
Mortality in children aged 12-59 month | 3-month time interval (total of 8 intervals per cluster)
  Mortality rate (deaths per 1000 years at risk) among children who were 12-59 month old when the latest azithromycin MDA took place in their village of residence.
Percentage of guardians and health care workers reporting MDA acceptable | 24 months after enrollment
  Data collected through interviews of guardians and health care workers to assess acceptability of MDA.
Percentage of the study population reached with MDA | 24 months after enrollment
  Data collected on MDA distribution and through interviews of guardians and health care workers to assess equity of MDA.
Cost and Cost-effectiveness of the intervention | 24 months after enrollment
  Data collected on MDA distribution to assess the economic aspects of MDA.The effectiveness will be determined by the trial outcome - both the primary outcome of mortality and the secondary outcomes of morbidity and possible AMR effects. The effectiveness will be expressed in different units such as deaths averted, or disability adjusted life years (DALYs).

CONTACTS AND LOCATIONS:
Overall Officials: Per Ashorn, MD, PhD, Principal Investigator — Center for Child Health Research, Tampere University; Ulla Ashorn, PhD, Principal Investigator — Center for Child Health Research, Tampere University; Samba Sow, MD, MSc, Principal Investigator — Center for Vaccine Development CVD-Mali; Nigel Klein, MBBS, PhD, Principal Investigator — University College London Hospitals; Camilla Ducker, MBBS, MSc, Principal Investigator — Tro Da Ltd, UK; Yin Bun Cheung, PhD, Principal Investigator — Centre for Quantitative Medicine, Duke-NUS Medical School; Dagmar Alber, PhD, Principal Investigator — University College London Hospitals
Locations (1):
- Center for Vaccine Development CVD-Mali, Bamako, Mali

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the trial, after deidentification. (The details are to be determined).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting 6 months after publication
Access Criteria: (The details are to be determined)

REFERENCES:
- [Derived] Haidara FC, Adubra L, Abdou M, Alber D, Ashorn U, Cheung YB, Cloutman-Green E, Diallo M, Ducker C, Fan YM, Gruffudd G, Hallamaa L, Haapaniemi T, Ihamuotila R, Juma J, Klein N, Luoma J, Martell O, Murugesan A, Okello C, Samake O, Traore CAT, Vehmasto T, Ylikruuvi K, Sow S, Ashorn P. Mass Administration of Azithromycin to Infants in Mali to Reduce Mortality. N Engl J Med. 2025 Oct 16;393(15):1498-1508. doi: 10.1056/NEJMoa2504644. PMID 41092331
- [Derived] Luoma J, Adubra L, Alber D, Ashorn P, Ashorn U, Cloutman-Green E, Diallo F, Ducker C, Elovainio R, Fan YM, Gates L, Gruffudd G, Haapaniemi T, Haidara F, Hallamaa L, Ihamuotila R, Klein N, Martell O, Sow S, Vehmasto T, Cheung YB. Statistical analysis plan for the LAKANA trial: a cluster-randomized, placebo-controlled, double-blinded, parallel group, three-arm clinical trial testing the effects of mass drug administration of azithromycin on mortality and other outcomes among 1-11-month-old infants in Mali. Trials. 2023 Nov 15;24(1):733. doi: 10.1186/s13063-023-07771-6. PMID 37968741
- [Derived] Adubra L, Alber D, Ashorn P, Ashorn U, Cheung YB, Cloutman-Green E, Diallo F, Ducker C, Elovainio R, Fan YM, Gates L, Gruffudd G, Haapaniemi T, Haidara F, Hallamaa L, Ihamuotila R, Klein N, Luoma J, Martell O, Sow S, Vehmasto T; LAKANA Trial Team. Testing the effects of mass drug administration of azithromycin on mortality and other outcomes among 1-11-month-old infants in Mali (LAKANA): study protocol for a cluster-randomized, placebo-controlled, double-blinded, parallel-group, three-arm clinical trial. Trials. 2023 Jan 3;24(1):5. doi: 10.1186/s13063-022-06966-7. PMID 36597115
- See also: The study website providing access to essential study materials, including the study protocol, Statistical Analysis Plan (SAP), Standard Operating Procedures (SOPs), and Data Collection Forms (DCFs). — https://lakana.org/

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-11-13): https://cdn.clinicaltrials.gov/large-docs/11/NCT04424511/Prot_SAP_ICF_002.pdf